CLINICAL TRIAL: NCT03489785
Title: Predictive Factors of Unpredicted Movement in Motor Evoked Potential During Intraoperative Neurophysiologic Monitoring in Adult Patients Undergoing Brain Surgery.
Brief Title: Predictive Factors of Unpredicted Movement in Motor Evoked Potential
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-1801-444-102
Record Dates: First submitted 2018-03-07; First posted 2018-04-05 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-01

CONDITIONS: Involuntary Movements; Brain Surgery
Keywords: Predicted factor; Motor Evoked Potentials
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Movement: If there is unexpected movement
- No movement: If there is no unexpected movement

SUMMARY:
The purpose of this study was to identify the predictive factors of unpredicted movement in motor evoked potential (MEP) during intraoperative neurophysiologic monitoring in adult patients undergoing brain surgery.

DETAILED DESCRIPTION:
Despite advances in neuroendovascular techniques, several complications can occur by brain urgery. Therefore, for neurosurgeons and anesthesiologists, it is a major concern to describe and monitor surgical lesion for maintaining structural and functional integrity as well as achieving maximal cytoreduction in lesion, and modifying the management of patients on the process of surgery. For example, microvascular Doppler sonography, indocyanine green aniography, intraoperative digital subtraction angiography, and intraoperative neurophysiologic monitoring (IONM) are used for this purpose.

The incidence of unpredictable and unacceptable movement is relative low. However, the results are so horrendous that they can cause injuries in site of rigid pin fixation of the head, cervical spine injuries, excessive surgical field movement, and deterioration of surgical outcome. However, risk factors associated with unpredictable and unacceptable movement remain unclear. Therefore, the aim of this retrospective study was to evaluate risk factors associated with unpredictable and unacceptable movement in the patients who underwent brain surgery with MEP monitoring under general anesthesia while using neuromuscular blocking agent.

The investigators recorded demographic data including age in years, sex, height in meters, weight in kilograms, body mass index (BMI in kg/m^2), ASA physical status class, diagnosed disease, performed surgical procedure, duration of anesthesia in minutes, duration of surgery in minutes, underlying disease (e.g. hypertension, diabetes, neurologic disease, respiratory disease), medications. Laboratory data was also collected including arterial blood gas analysis, hematocrit, hemoglobin, sodium, potassium, ionized calcium, ionized magnesium, and lactate. Unpredictable and unacceptable movement was defined as either the dangerous gross movement requiring the increase the continuous infusion rate of rocuronium in view of the surgeon, anesthesiologist, and neurophysiologic specialist or the shake of the surgical field requiring the increase the continuous infusion rate of rocuronium.

ELIGIBILITY:
Inclusion Criteria:

* From June 2003 to August 2017, patients who underwent motor-evoked potential monitoring during brain surgery under partial neuromuscular relaxation at the Seoul National University Bundang Hospital.

Exclusion Criteria:

* Age : 18 or younger and 75 or older
* Anesthesiologists physical status classes III or more
* body mass index(BMI) < 18.5 kg/m^2 or BMI > 25 kg/m^2
* Patients who received medications that affect muscle relaxation recovery other than anticonvulsants
* OT/PT > 40 IU/L, Cr > 1.4 mg/dl
* Moderate to severe respiratory or heart disease

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From June 2003 to August 2017, patients who underwent motor-evoked potential monitoring during brain surgery under partial neuromuscular relaxation at the Seoul National University Bundang Hospital were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2003-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive factors of unpredicted movement | during brain surgery
  The investigators retrospectively compare the data of patients with and without unpredictable and unacceptable movement during surgery. For continuous variables, values were compared using the independent t-test. Differences in proportions were compared using chi-square test. Variables with P-values < 0.05 in the primary test were selected and univariate binary logistic regression analyses were conducted to identify the factors predictive of an unpredictable and unacceptable movement. P-value < 0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided